CLINICAL TRIAL: NCT02219399
Title: Maternal DHA Supplementation and Pregnancy Outcome
Brief Title: DHA Supplementation and Pregnancy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 00186H
Record Dates: First submitted 2014-06-09; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Pregnancy
Keywords: Pregnancy; DHA; Gestational Length; Cognitive Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 300 mg DHA (Experimental): 300 mg DHA
  Interventions: Dietary Supplement: 300 mg DHA
- Placebo (Placebo Comparator): olive oil or high oleic acid sunflower oil placebo
  Interventions: Dietary Supplement: Placebo
- 600 mg DHA (Experimental): 600 mg DHA
  Interventions: Dietary Supplement: 600 mg DHA

INTERVENTIONS:
Dietary Supplement: 600 mg DHA — Pregnant women were given 600 mg DHA in the last trimester of pregnancy
  Arms: 600 mg DHA
Dietary Supplement: 300 mg DHA — Pregnant women were given 300 mg DHA in the last trimester of pregnancy and through the first 3 months of breastfeeding
  Arms: 300 mg DHA
Dietary Supplement: Placebo — Pregnant women in the control group received placebo of either olive oil or high oleic acid sunflower oil during the study period
  Arms: Placebo

SUMMARY:
Supplementation with DHA during pregnancy will increase gestational length and improve cognitive development.

DETAILED DESCRIPTION:
This was a trial of supplementation with DHA during pregnancy to increase gestational length. Subjects were provided with 300 mg, 600 mg or placebo (olive oil) in a randomized design from week 24-26 of pregnancy until delivery. Gestational age, birth weight and birth length data were collected and infants growth at 2 and 4 months and cognitive development at 4 months and 1 year were measured.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* 18 years of age or older

Exclusion Criteria:

* cervical incompetence
* presence of cervical cerclage
* placenta previa
* intrauterine infection
* known substance abuse
* multiple fetuses
* current pre-eclampsia
* preexisting diabetes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 871 (Actual)
Dates: Start 2001-01; Primary Completion 2004-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Gestational Length | 13 weeks
  Length of gestation as measured by Last menstrual period method and US
Cognitive Development | 4 months
  Bayley's Scales of Infant Development measured at 4 months of age
Cognitive Development | 12 months
  Bayley's Scales of Infant Development measured at 12 months of age

SECONDARY OUTCOMES:
Infant birth length | 13 weeks
  self-explanatory
Infant Growth Velocity | 2 months to 4 months of age
  Change in infant length and weight from 2 to 4 months of age
Infant birth weight | 13 weeks
  self-explanatory
Infant head circumference at birth | 13 weeks
  self-explanatory

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Harris, PhD, Principal Investigator — Colorado State University
Locations (2):
- United States (2):
  - Denver Health Hospitals and Clinics, Denver, Colorado
  - Colorado State University, Fort Collins, Colorado